CLINICAL TRIAL: NCT01560234
Title: A Double-blind, Placebo-controlled, Randomised Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Inhaled Doses of AZD8848 in Healthy Subjects
Brief Title: AZD8848 Single Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D0542C00001; Eudract number 2011-005986-20
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Safety; tolerability; healthy; pharmacokinetic; pharmacodynamic; inhaled
MeSH Terms: conditions — Respiratory Aspiration | interventions — AZD8848

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- AZD8848 (Experimental)
  Interventions: Drug: AZD8848
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD8848 — Single dose, oral inhalation (nebuliser solution)
  Arms: AZD8848
Drug: Placebo — Single dose, oral inhalation (nebuliser solution)
  Arms: Placebo

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single ascending doses of AZD8848 in healthy subjects.

DETAILED DESCRIPTION:
A Double-blind, Placebo-controlled, Randomised Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Inhaled Doses of AZD8848 in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or women aged 18 to 45 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
* Women can be of childbearing potential and must have been stable on a highly effective contraceptive method for at least 3 months prior to Visit 1 (screening) and be willing to continue on the chosen contraceptive method
* Male subjects should be willing to use a condom (with spermicide) to prevent pregnancy and drug exposure of a female partner and refrain from donating sperm or fathering a child from the day of the investigational product administration until 3 months
* Have a body mass index (BMI) between 18 and 30 kg/m2 and weigh at least 50 kg and no more than 100 kg
* Ability to produce sputum of good enough quality for assessment of biomarkers

Exclusion Criteria:

* Abnormal vital signs, after 10 minutes supine rest, defined as any of the following (SBP > 140 mmHg, Diastolic blood pressure (DBP) > 90 mmHg, Heart rate < 40 or > 85 beats per minute)
* Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome
* History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class as AZD8848
* History of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT syndrome, or sudden death)
* History of asthma or allergic rhinitis

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Aggarwal, Study Director — AstraZeneca R&D, 35 Gatehouse Drive, MA 02451 USA; James Ritter, BA,MA D Phil,BM BCh,MRCP,FRCP, Principal Investigator — Quintile Drug Research Unit at Guy's Hospital Quintiles Ltd 6 Newcomen Street London SE1 1YR United Kingdom
Locations (1):
- Research Site, London, United Kingdom

REFERENCES:
- [Derived] Delaney S, Biffen M, Maltby J, Bell J, Asimus S, Aggarwal A, Kraan M, Keeling D. Tolerability in man following inhalation dosing of the selective TLR7 agonist, AZD8848. BMJ Open Respir Res. 2016 Feb 23;3(1):e000113. doi: 10.1136/bmjresp-2015-000113. eCollection 2016. PMID 26933507
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1660&filename=D0542C00001_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 47 male and female subjects (6 cohorts with additional 2 cohorts) were randomized in the study.There were 6 subjects per cohort (4 subjects received AZD8848 and 2 subjects received placebo), with the exception of Cohort 3 (1.5 μg), where 3 subjects received AZD8848 and 2 subjects received placebo.
Groups:
- Placebo: Commercial 0.9% sodium chloride solution.
- Cohort 1: AZD8848 0.15 μg
- Cohort 2: AZD8848 0.5 ug
- Cohort 3: AZD8848 1.5 μg
- Cohort 4: AZD8848 5 μg
- Cohort 5: AZD8848 15 μg
- Cohort 7: AZD8848 15 μg (Multiple Inhalation)
- Cohort 6 and 8: AZD8848 30 μg (similar investigational product administration conditions)
Period: Overall Study
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Started | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8
Completed | 13 | 4 | 3 | 3 | 4 | 2 | 4 | 6
Not Completed | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 2
Not completed — Lost to Follow-up | 3 | 0 | 1 | 0 | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All available data were used for the baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8 | Total
Number analyzed (Participants) | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8 | 47
Age, Continuous [Mean (Standard Deviation); unit: Years] | 27 (6) | 29 (10) | 23 (3) | 24 (5) | 31 (4) | 27 (6) | 30 (9) | 31 (9) | 28 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 2 | 2 | 4 | 2 | 3 | 1 | 23
  Male | 8 | 3 | 2 | 1 | 0 | 2 | 1 | 7 | 24
Subject characteristics (Height) [Mean (Standard Deviation); unit: cm] | 170.1 (7.1) | 168.6 (1.7) | 170.5 (8.5) | 167.7 (15.5) | 166.0 (5.0) | 175.0 (8.3) | 169.3 (11.1) | 176.9 (8.6) | 170.9 (8.3)
Subject characteristics (Weight) [Mean (Standard Deviation); unit: kg] | 72.1 (11.2) | 76.9 (6.7) | 68.2 (12.2) | 71.4 (5.0) | 67.7 (14.2) | 78.1 (16.3) | 69.4 (10.5) | 79.3 (8.0) | 73.3 (10.9)
Subject characteristics (BMI) [Mean (Standard Deviation); unit: kg/m²] | 24.81 (2.71) | 27.02 (1.94) | 23.41 (3.50) | 25.63 (3.16) | 24.48 (4.46) | 25.31 (3.47) | 24.41 (4.87) | 25.40 (2.37) | 25.01 (3.00)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Summary of number of subjects who had at least one adverse event
Time Frame: Screening up to Day 13
Population: Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8
participants | 6 | 2 | 1 | 0 | 3 | 1 | 2 | 4

2. Secondary Outcome: Summary (Geometric Mean and GCV%) of Pharmacokinetic Parameters of Total AZ12432045 - AUC (Nmol*h/L)
Time Frame: On Day 1 at 0min, 2min, 5min, 10min, 20min, 30min, 45min, 60min, 90min, 2h, 4h, 6h, 8h, 12h, 24h and 48h
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 5
nmol*h/L |  |  |  |  | 0.149 (22.9) | 0.360 (43.4) | 0.312 (26.2) | 0.642 (21.9)
Statistical Analysis 1: Comparison: Cohort 4 vs Cohort 5 vs Cohort 7 vs Cohort 6 and 8; Test type: Superiority or Other; Regression, Linear; Slope = 0.81, 90% CI 2-sided [0.63 to 1.00], Standard Error of Mean 0.10 — AUC (nmol*h/L) 5 to 30 μg

3. Secondary Outcome: Summary (Geometric Mean and GCV%) of Pharmacokinetic Parameters of Total AZ12432045 - AUC(0-t) (Nmol*h/L)
Time Frame: On Day 1 at 0min, 2min, 5min, 10min, 20min, 30min, 45min, 60min, 90min, 2h, 4h, 6h, 8h, 12h, 24h and 48h
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 5
nmol*h/L |  |  |  |  | 0.131 (22.1) | 0.328 (46.2) | 0.279 (26.6) | 0.591 (22.3)
Statistical Analysis 1: Comparison: Cohort 4 vs Cohort 5 vs Cohort 7 vs Cohort 6 and 8; Test type: Superiority or Other; Regression, Linear; Slope = 0.84, 90% CI 2-sided [0.65 to 1.04], Standard Error of Mean 0.11 — AUC(0-t) (nmol*h/L) 5 to 30 μg

4. Secondary Outcome: Summary (Geometric Mean and GCV%) of Pharmacokinetic Parameters of Total AZ12432045 - Cmax (Nmol/L)
Time Frame: On Day 1 at 0min, 2min, 5min, 10min, 20min, 30min, 45min, 60min, 90min, 2h, 4h, 6h, 8h, 12h, 24h and 48h
Population: Pharmacokinetic Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 0 | 0 | 4 | 3 | 4 | 4 | 4 | 5
nmol/L |  |  | 0.0362 (10.3) | 0.0903 (40.8) | 0.473 (36.1) | 0.963 (47.0) | 0.629 (13.6) | 1.67 (18.6)
Statistical Analysis 1: Comparison: Cohort 2 vs Cohort 3 vs Cohort 4 vs Cohort 5 vs Cohort 7 vs Cohort 6 and 8; Test type: Superiority or Other; Regression, Linear; Slope = 0.95, 90% CI 2-sided [0.87 to 1.04], Standard Error of Mean 0.05 — Cmax (nmol/L) 0.5 to 30 μg

5. Secondary Outcome: Statistical Assessment of CXCL10 Ratio-to-baseline - Plasma
Description: Smmarizes the statistical assessment comparing active CXCL10 ratio to baseline to placebo at each dose level, sampling time, and matrix
Time Frame: Baseline, 24 Hours.
Population: Pharmacodynamic Population Set
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8
ratio | 0.9290 (10.4) [0.7703 to 1.120] | 0.9267 (107.7) [0.6381 to 1.346] | 0.8638 [0.5949 to 1.254] | 0.9869 [0.6417 to 1.518] | 1.355 [0.9332 to 1.967] | 2.079 [1.412 to 3.059] | 2.120 [1.460 to 3.078] | 6.354 [4.880 to 8.274]
Statistical Analysis 1: Comparison: Placebo vs Cohort 1; 24 hour Plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 99.75, 95% CI 2-sided [65.76 to 151.32] — Cohort 1/0.15 ug vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cohort 2; 24 hour Plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 92.99, 95% CI 2-sided [61.21 to 141.27] — Cohort 2/1.5ug vs Placebo
Statistical Analysis 3: Comparison: Placebo vs Cohort 4; 24 hour Plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 145.83, 95% CI 2-sided [96.11 to 221.28] — Cohort 4/5 ug vs Placebo
Statistical Analysis 4: Comparison: Placebo vs Cohort 3; 24 hour Plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 106.23, 95% CI 2-sided [66.42 to 169.93] — Cohort 3/1.5 ug vs Placebo
Statistical Analysis 5: Comparison: Placebo vs Cohort 5; 24 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 223.76, 95% CI [144.98 to 345.35] — Cohort 5/15 μg vs Placebo
Statistical Analysis 6: Comparison: Placebo vs Cohort 7; 24 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 228.23, 95% CI 2-sided [150.36 to 346.41] — Cohort 7/15 μg vs Placebo
Statistical Analysis 7: Comparison: Placebo vs Cohort 6 and 8; 24 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 684.03, 95% CI 2-sided [495.31 to 944.65] — Cohort 6 and 8/30 μg vs Placebo

6. Secondary Outcome: Statistical Assessment of CXCL10 Ratio-to-baseline - Plasma
Description: Smmarize the statistical assessment comparing active CXCL10 ratio to baseline to placebo at each dose level, sampling time, and matrix
Time Frame: Baseline, 48 Hours
Population: Pharmacodynamic Population Set
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8
ratio | 1.009 (10.4) [0.8914 to 1.142] | 0.9669 (107.7) [0.7552 to 1.238] | 0.9256 [0.7229 to 1.185] | 1.134 [0.8524 to 1.508] | 1.211 [0.9460 to 1.550] | 1.036 [0.8020 to 1.338] | 1.482 [1.158 to 1.897] | 2.422 [2.034 to 2.885]
Statistical Analysis 1: Comparison: Placebo vs Cohort 1; 48 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 95.81, 95% CI 2-sided [72.70 to 126.28] — Cohort 1/0.15 ug vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cohort 2; 48 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 91.72, 95% CI 2-sided [69.53 to 121.00] — Cohort 2/0.5 ug vs Placebo
Statistical Analysis 3: Comparison: Placebo vs Cohort 3; 48 hour Plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 112.34, 95% CI 2-sided [82.30 to 153.35] — Cohort 3/1.5 ug vs Placebo
Statistical Analysis 4: Comparison: Placebo vs Cohort 4; 48 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 120.00, 95% CI 2-sided [91.04 to 158.18] — Cohort 4/5 ug vs Placebo
Statistical Analysis 5: Comparison: Placebo vs Cohort 5; 48 hour placebo; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 102.67, 95% CI 2-sided [77.02 to 136.87] — Cohort 5/15 ug vs Placebo
Statistical Analysis 6: Comparison: Placebo vs Cohort 7; 48 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 146.86, 95% CI 2-sided [111.39 to 193.62] — Cohort 7/15 ug vs Placebo
Statistical Analysis 7: Comparison: Placebo vs Cohort 1; 48 hour plasma; Test type: Superiority or Other; ANCOVA; Percentage of Placebo = 240.04, 95% CI 2-sided [193.82 to 297.28] — Cohort 6 and 8/30 ug

7. Primary Outcome: Summary for Lymphocytes Laboratory Results
Time Frame: Baseline, Day 1, Day 2, Day 3, and Follow up (up to Day 13)
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8
cells*10^9/L
  Baseline | 1.6 (0.3) | 1.7 (0.5) | 2.0 (0.6) | 2.1 (0.5) | 2.3 (0.7) | 2.1 (0.3) | 1.9 (0.3) | 1.6 (0.3)
  Day 1 | 2.3 (0.5) | 2.1 (0.7) | 2.7 (0.7) | 2.2 (0.3) | 2.4 (0.6) | 2.4 (0.6) | 2.0 (0.4) | 1.4 (0.6)
  Day 2 | 1.6 (0.4) | 2.0 (0.6) | 1.9 (0.3) | 2.0 (1.5) | 2.2 (0.7) | 2.0 (0.3) | 1.4 (0.3) | 0.9 (0.2)
  Day 3 | 1.8 (0.5) | 2.0 (0.6) | 2.1 (0.2) | 2.0 (0.6) | 2.3 (1.0) | 2.0 (0.1) | 1.7 (0.1) | 1.4 (0.2)
  Follow up (up to Day 13) | 1.7 (0.4) | 2.0 (0.5) | 2.1 (0.5) | 1.8 (0.3) | 2.1 (0.8) | 1.9 (0.2) | 1.7 (0.3) | 1.5 (0.4)

8. Secondary Outcome: Statistical Assessment of CXCL10 Ratio-to-baseline- Sputum
Description: Summarize the statistical assessment comparing active CXCL10 ratio to baseline to placebo at each dose level, sampling time, and matrix
Time Frame: Baseline, 24 Hours.
Population: Pharmacodynamic Population Set
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Number analyzed (Participants) | 16 | 4 | 4 | 3 | 4 | 4 | 4 | 8
ratio | 1.038 (10.4) [0.5929 to 1.818] | 1.192 (107.7) [0.4145 to 3.430] | 0.8500 [0.2976 to 2.428] | 0.8465 [0.2396 to 2.991] | 3.160 [0.9011 to 11.08] | 2.012 [0.7055 to 5.737] | 4.858 [1.704 to 13.85] | 11.29 [3.792 to 33.60]
Statistical Analysis 1: Comparison: Placebo vs Cohort 1; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 114.87, 95% CI 2-sided [34.83 to 378.78] — Cohort 1/0.15 ug vs Placebo
Statistical Analysis 2: Comparison: Placebo vs Cohort 2; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 81.89, 95% CI 2-sided [24.96 to 268.70] — Cohort 2/0.5 ug vs Placebo
Statistical Analysis 3: Comparison: Placebo vs Cohort 3; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 81.55, 95% CI 2-sided [20.63 to 322.42] — Cohort 3/1.5 ug vs Placebo
Statistical Analysis 4: Comparison: Placebo vs Cohort 4; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 304.37, 95% CI 2-sided [76.61 to 1209.33] — Cohort 4/5 ug vs Placebo
Statistical Analysis 5: Comparison: Placebo vs Cohort 5; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 193.80, 95% CI 2-sided [59.01 to 636.49] — Cohort 5/15 μg vs Placebo
Statistical Analysis 6: Comparison: Placebo vs Cohort 7; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 467.96, 95% CI 2-sided [142.77 to 1533.92] — Cohort 7/15 μg vs Placebo
Statistical Analysis 7: Comparison: Placebo vs Cohort 6 and 8; 24 hour Sputum; Test type: Superiority or Other; ANCOVA; Comparison of Placebo = 1087.35, 95% CI 2-sided [317.19 to 3727.57] — Cohort 6 and 8/30 μg vs Placebo

ADVERSE EVENTS:
Time Frame: Screening up to 11 - 13 Months
Arm/Group | Placebo | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Cohort 7 | Cohort 6 and 8
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/4 | 0/4 | 0/3 | 1/4 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 6/16 | 2/4 | 1/4 | 0/3 | 3/4 | 1/4 | 2/4 | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=16) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=3) | Cohort 4 (N=4) | Cohort 5 (N=4) | Cohort 7 (N=4) | Cohort 6 and 8 (N=4)
Pelvic Inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=16) | Cohort 1 (N=4) | Cohort 2 (N=4) | Cohort 3 (N=3) | Cohort 4 (N=4) | Cohort 5 (N=4) | Cohort 7 (N=4) | Cohort 6 and 8 (N=8)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0/4 (0)
chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a publication (e.g., in a scientific journal) based on the results of this study is envisaged, approval from AstraZeneca will be obtained and a draft manuscript will be submitted to AstraZeneca for scrutiny and comment. The choice of conduit will be mutually agreed on by the Principal Investigator and AstraZeneca.